CLINICAL TRIAL: NCT05678413
Title: Role of Paclitaxel in Prevention of Stricture Recurrence After Direct Visual Internal Urethrotomy (DVIU); Prospective Clinical Trial
Brief Title: Role of Paclitaxel in Stricture Urethra
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Intraurethral Paclitaxel
Record Dates: First submitted 2022-12-24; First posted 2023-01-10 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Stricture Urethra
Keywords: DVIU, Stricture, Paclitaxel
MeSH Terms: conditions — Urethral Stricture; Constriction, Pathologic | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: Cystourethroscopy will be performed using a 22 Fr rigid cystoscope to allow for ureteric catheter 3F/a wire to be passed through the stricture and into the urinary bladder. DVIU will be performed by cold-knife incisions at the 12-, 3-, and 9 o'clock positions through the full thickness of the fibrosis to healthier appearing tissue. A 23 Fr Wolf (Vernon Hills, IL) injection scope and a standard injection needle was used to inject 30 mg/5mL of paclitaxel vial, 1.5 mL will be injected along the length of each incision into healthier appearing tissue for a total of 5 mL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DVIU with paclitaxel (Active Comparator): Cystourethroscopy will be performed using a 22 Fr rigid cystoscope to allow for ureteric catheter 3F/a wire to be passed through the stricture and into the urinary bladder. DVIU will be performed by cold-knife incisions at the 12-, 3-, and 9 o'clock positions through the full thickness of the fibrosis to healthier appearing tissue. A 23 Fr Wolf (Vernon Hills, IL) injection scope and a standard injection needle was used to inject 30 mg/5mL of paclitaxel vial, 1.5 mL will be injected along the length of each incision into healthier appearing tissue for a total of 5 mL.
  Interventions: Procedure: DVIU with paclitaxel injection
- DVIU (Active Comparator): Cystourethroscopy will be performed using a 22 Fr rigid cystoscope to allow for ureteric catheter 3F/a wire to be passed through the stricture and into the urinary bladder. DVIU will be performed by cold-knife incisions at the 12-, 3-, and 9 o'clock positions through the full thickness of the fibrosis to healthier appearing tissue.
  Interventions: Procedure: DVIU

INTERVENTIONS:
Procedure: DVIU with paclitaxel injection — Cystourethroscopy will be performed using a 22 Fr rigid cystoscope to allow for ureteric catheter 3F/a wire to be passed through the stricture and into the urinary bladder. DVIU will be performed by cold-knife incisions at the 12-, 3-, and 9 o'clock positions through the full thickness of the fibrosis to healthier appearing tissue. A 23 Fr Wolf (Vernon Hills, IL) injection scope and a standard injection needle was used to inject 30 mg/5mL of paclitaxel vial, 1.5 mL will be injected along the length of each incision into healthier appearing tissue for a total of 5 mL.
  Arms: DVIU with paclitaxel
Procedure: DVIU — DVIU
  Arms: DVIU

SUMMARY:
Stricture urethra is a common disease and has various causing factors. The most common performed procedure is direct visual internal urethrotomy (DVIU), but unfortunately has a high recurrence rates. Multiple trial were performed to improve the outcomes of DVIU. Various intralesional injections were used. in this trial we will evaluate intralesional paclitaxel injection following DVIU.

ELIGIBILITY:
Inclusion Criteria:

* Anterior urethral stricture
* Short strictures (less than 2 cm)
* International Prostate Symptom Score less than 11 and maximum flow rate < 15 ml per second.
* No previous treatment for stricture disease

Exclusion Criteria:

* Recurrent cases
* Prior pelvic radiation
* Associated other pathology or unresolved confounding etiologies (e.g. bladder neck contracture, neurogenic bladder, benign prostatic hyperplasia) were excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Success of treatment | 1 year
  Treatment free rates (Freedom from repeat intervention e.g., repeat dilation, DVIU or urethroplasty).

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Fawzy Salman, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided